CLINICAL TRIAL: NCT04714281
Title: Comparison of Clinical Performance and Hemocompatibility of Dialyzers Applied During Post-dilution Online Hemodiafiltration - eMPORA III Study (Modified POlysulfone membRAne)
Brief Title: Comparison of Clinical Performance and Hemocompatibility of Dialyzers Applied During Post-dilution Online Hemodiafiltration
Acronym: eMPORAIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Institut Dr. Schauerte GmbH (IDS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HD-FX-08-EU; CIV-20-10-035024 (Other: EUDAMED)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Renal Failure; End Stage Renal Disease
Keywords: Hemodialysis; Hemodiafiltration; Renal replacement therapy; Dialyzer
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Kidneys, Artificial

STUDY DESIGN:
Intervention Model Description: Prospective, open, controlled, cross-over (with randomized treatment sequences), interventional, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodiafiltration HDF (Other): Three consecutive treatment periods of four weeks, one last study week where the patient is re-assigned to the same type of dialyzer used before beginning the study and one follow-up week per patient. Each treatment period includes 12 hemodiafiltration HDF sessions and is assigned to one type of dialyzer: FX CorAL 600 Fresenius Medical Care, comparator FX CorDiax 600 Fresenius Medical Care and comparator xevonta Hi 15 (B. Braun).
  Interventions: Device: Dialyser

INTERVENTIONS:
Device: Dialyser — Three consecutive treatment periods of four weeks, one last study week where the patient is re-assigned to the same type of dialyzer used before beginning the study and one follow-up week per patient. Each treatment period includes 12 hemodiafiltration HDF sessions and is assigned to one type of dialyzer: FX CorAL 600 Fresenius Medical Care, comparator FX CorDiax 600 Fresenius Medical Care and comparator xevonta Hi 15 (B. Braun).

SUMMARY:
Comparison of the clinical performance and the hemocompatibility profile of different high-flux dialyzers, all applied during post-dilution online hemodiafiltration

DETAILED DESCRIPTION:
The primary objective of this study is to test whether the hemodialyzer FX CorAL 600 (applied during post-dilution online hemodiafiltration) is non-inferior or superior to the comparator hemodialyzers FX CorDiax 600 and xevonta Hi 15 in removing ß2-microglobulin.

The secondary objectives of this study are:

* To compare the FX CorAL 600 dialyzer with the comparator hemodialyzers FX CorDiax 600 and xevonta Hi 15 regarding their efficacies in removing other uremic toxins.
* To compare the FX CorAL 600 dialyzer with the comparator hemodialyzers FX CorDiax 600 and xevonta Hi 15 regarding their hemocompatibility profiles.

ELIGIBILITY:
Inclusion Criteria:

General:

* Minimum age of 18 years
* Existing informed consent form signed and dated by study patient as well as investigator/authorized physician
* The patient is legally competent and able to understand the nature, risks, meaning, and consequences of the clinical trial and can subsequently declare her/his consent for participation in the clinical trial (cf. European Medical Device Directive and corresponding national regulations)
* Patients with a chronic kidney disease stage 5D (end stage renal disease with a glomerular filtration rate of 15 ml/min or less) on hemodiafiltration as extracorporeal renal replacement therapy

Study-specific:

* On online post-dilution hemodiafiltration (HDF), at least 4 h treatment time thrice weekly with FX or FX CorDiax dialyzer ≥ 1 month
* Vascular access (fistula or graft) which enables blood flow rate ≥ 300 ml/min

Exclusion Criteria:

General:

* Any condition which could interfere with the patient's ability to comply with the study. This decision is at the discretion of the treating physician and relates to the general stable condition of the patient (e.g. any acute condition, e.g. infection or mental problem which might give reason for concern etc.)
* Ongoing participation in an interventional clinical study during the preceding 30 days
* Previous participation in this study
* Pregnancy (pregnancy test will be conducted at start and end of study with female patients aged < 55 years) or lactation period
* Patient is not able to give informed consent according to the European Medical Device Directive and corresponding national regulations

Study-specific:

* Recurrent episodes of vascular access failure characterized by e.g. repeated cannulation problems or unstable blood flows within the last 2 months prior to study start (>3 times, respectively)
* Repeated single needle treatments (>3 times within the last 2 months prior to study start)
* Catheter as vascular access
* Unstable patients (due to e.g. acute intercurrent disease like cardiovascular infarction, decompensated heart failure, cerebrovascular accident, severe infection, active malignant disease)
* Patients with NYHA ≥ 3, COPD (GOLD 2-4), frequent intradialytic symptomatic hypotension
* Patients with known or suspected allergy to trial product and related products
* Patients with known inborn or acquired deficiencies of the innate and/or adaptive immune system
* Patients with acute (use within last 4 weeks) and/or chronic immunosuppressive medication e.g. due to immune-mediated disease including autoimmune diseases, transplantation, or cancer (oral and systemic corticosteroids, calcineurin and mTOR-inhibitors, immunosuppressive monoclonal antibodies, cytotoxic chemotherapy)
* Planned absence from dialysis unit within the 14 weeks of study duration e.g. due to scheduled hospitalization, holidays or any other reason
* Active HBV, HCV, HIV, SARS-CoV-2 infection, as well as any other febrile illness
* Reported SARS-CoV-2 infection with or without symptoms within the 12 weeks before inclusion into the study
* Unwillingness to undergo repeated SARS-CoV-2 infection testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Removal rate of β2-microglobulin | t=240 minutes of HDF
  Removal rate of β2-microglobulin will be calculated a primary endpoint in blood samples to evaluate the clinical Performance of the dialyzer FXCorAL

CONTACTS AND LOCATIONS:
Overall Officials: Götz Ehlerding, Dr med, Principal Investigator — Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen
Locations (8):
- Czechia (2):
  - Fresenius Nephrocare Nymburk, Nymburk
  - Fresenius Nephrocare Praha 9 - Vysocany, Prague
- Germany (4):
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - PHV-Dialysezentrum Goslar, Goslar
  - Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen, Hanover
  - PHV Dialysezentrum Kiel, Kiel
- Hungary (2):
  - Péterfy II. Dialízis Központ, Budapest
  - Váci Dialízis Központ, Vác

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ehlerding G, Ries W, Kempkes-Koch M, Ziegler E, Ronova P, Krizsan M, Veresova J, Boke M, Erlenkotter A, Nitschel R, Zawada AM, Kennedy JP, Braun J, Larkin JW, Korolev N, Lang T, Ottillinger B, Stauss-Grabo M, Griesshaber B. Randomized investigation of increased dialyzer membrane hydrophilicity on hemocompatibility and performance. BMC Nephrol. 2024 Jul 10;25(1):220. doi: 10.1186/s12882-024-03644-5. PMID 38987671
- See also: Link to PubMed ID 38987671 — https://pubmed.ncbi.nlm.nih.gov/38987671/